CLINICAL TRIAL: NCT02388126
Title: Prostate Magnetic Resonance Imaging in Patient With Previous Negative Biopsies
Acronym: PROMANEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Peter Boström, Adj. prof., Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T22/2015
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Experimental): Comparison of targeted transrectal ultrasound guided prostate biopsies based on 3T multiparametric MRI findings to systematic non-targeted transrectal ultrasound guided prostate biopsies
  Interventions: Device: 3T multiparametric MRI; Device: Transrectal ultrasound

INTERVENTIONS:
Device: 3T multiparametric MRI — Magnetom Verio 3T, Erlangen, Germany
Device: Transrectal ultrasound — Bk Medical Pro Focus Ultraview 2202 system

SUMMARY:
Prostate cancer has been the most common neoplastic disease in men in Finland over the last ten years. Prostate-specific antigen (PSA) plays an important role in screening of prostate cancer. However, PSA has a limited sensitivity and specificity for prostate cancer detection. Commonly, the diagnosis of prostate cancer is done by transrectal ultrasonography (TRUS) guided biopsy. Because of the low accuracy of TRUS a systematic biopsy is usually performed instead of targeted TRUS biopsy. While, as many as 47% of the ultra-sound guided biopsies may be false negative and biopsies carry a risk of increase in complications, there is an increasing interest in developing more accurate non-invasive imaging modalities.

This study will enroll 150 men with previous negative biopsies and clinical suspicion of prostate cancer due to serum level of PSA higher than 2.5 ng/ml or abnormal digital rectal examination (DRE) or patients in active surveillance due to low risk prostate carcinoma. Anatomical magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI) at 3 Tesla (T) magnetic field using surface coils will be used to non-invasively predict the presence or absence of prostate cancer. In addition to routine 12-core TRUS biopsies, targeted TRUS guided biopsy based on MRI findings will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Language spoken: Finnish or Swedish
* Clinical suspicion of prostate cancer and/or previous negative prostate biopsies and MRI target
* Previous diagnosis of prostate carcinoma and patient on active surveillance
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Language spoken: Finnish or Swedish
* Clinical suspicion of prostate cancer and/or previous negative prostate biopsies and MRI target
* Previous diagnosis of prostate carcinoma and patient on active surveillance
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of multiparametric MRI in prostate cancer diagnosis | 3 mounths
  Multiparametric MRI is performed in patients with previous negative biopsies with clinical suspicion of prostate cancer (elevated PSA and/or abnormal DRE) or in patients in active surveillance due to low risk prostate carcinoma. The accuracy will be determined using the results from transrectal ultrasound guided biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Boström, Adj. Prof., Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland